CLINICAL TRIAL: NCT03459391
Title: A Double-blind, Randomized, Placebo-controlled Study of the Safety,Tolerability and Pharmacokinetics of Increasing Doses of XC221 After Single and Repeated Oral Administration in Healthy Volunteers
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics of XC221 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ARI-XC221-01
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Influenza; Acute Respiratory Infection
Keywords: Healthy volunteers; Phase I; PHARMENTERPRISES
MeSH Terms: conditions — Influenza, Human | interventions — XC221

STUDY DESIGN:
Intervention Model Description: The dose cohorts were included into the study subsequently based on preliminary safety results evaluation performed by the Data Safety Monitoring Committee. 2 doses of XC221/placebo (60 mg and 200 mg) were used in the study.The duration of exposure to the study drug was 6 days in each cohort: Day 1, once, at the step of single administration, and then in 6 days, daily, 1 time a day for 5 days at the step of multiple administration.
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using Placebo equivalent to XC221 tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XC221 60 mg (Experimental): Cohort 1:16 subjects were randomized in a 3:1 ratio to be treated either with 60 mg XC221 (12 subjects) or placebo (4 subjects, see placebo arm).
  Interventions: Drug: XC221 60 mg
- XC221 200 mg (Experimental): Cohort 2: 16 subjects were randomized in a 3:1 ratio to be treated either with 200 mg XC221 (12 subjects) or placebo (4 subjects, see placebo arm).
  Interventions: Drug: XC221 200 mg
- Placebo (Placebo Comparator): Placebo comparator arm consists of 8 subjects (4 subjects from each cohort).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 60 mg — The volunteers received the study drug once, and then continued daily intake for 5 days after a 6-day break.
  Arms: XC221 60 mg
Drug: XC221 200 mg — The volunteers received the study drug once, and then continued daily intake for 5 days after a 6-day break.
  Arms: XC221 200 mg
Drug: Placebo — The volunteers received the study drug once, and then continued daily intake for 5 days after a 6-day break.
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety and tolerability of increasing doses of drug XC221 after single and repeated oral administration in healthy volunteers. The volunteers received the study drug once, and then continued daily intake for 5 days after a 6-day break. The primary objective of the study was to evaluate the safety and tolerability profile for drug XC221 after single and multiple administration based on the frequency and severity of adverse events and changes in vital signs, laboratory results, electrocardiography and results of the physical examination. The secondary objective of the study was to assess pharmacokinetics of active pharmaceutical substance XC221GI and its metabolite XC221A.

DETAILED DESCRIPTION:
One Russian center was approved for participation in this study. One center was initiated. Healthy volunteers were enrolled in 1 center. The study consisted of 4 periods: screening, single administration, multiple administration and follow-up.

All eligible subjects were randomized into the study in appropriate cohort groups sequentially. Cohort 1 - XC221 or Placebo 60 mg once and then daily 5 days after a 6-day break; Cohort 2 - XC221 or Placebo 200 mg once and then daily during 5 days after a 6-day break. The decision regarding increasing of the study drug dose for a subsequent cohort was made by the Data Safety Monitoring Committee on the basis of preliminary safety results assessment. A total of 24 volunteers received XC221 (60 mg or 200 mg) and a total of 8 volunteers received the placebo during the study participation. The follow-up period lasted for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking men aged 18 to 45 years (inclusive);
2. Verified diagnosis "healthy" according to standard clinical, laboratory and instrumental methods of examination;
3. Body mass >50 kg and body mass index of 18.5 to 30 kg/m2 (inclusive);
4. Negative result of tests for alcohol and drugs;
5. Consent to use reliable methods of contraception during the study and 3 months after its completion (condoms with spermicide);
6. Signed patient information sheet and informed consent form for participation in the study.

Exclusion Criteria:

1. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal system and also disease of digestive tract, liver, kidneys, blood;
2. Laboratory abnormalities at screening;
3. Surgical interventions on digestive tract in the anamnesis (except for an appendectomies);
4. Systolic pressure is less than 90 mm Hg. or more than 130 mm Hg., diastolic pressure is less than 60 mm Hg. or more than 85 mm Hg., pulse rate less than 60/min. or more than 80/min.;
5. Course intake of medicinal products (including herbs and biologically active additives) for preventive or curative purposes within 1 month prior to screening;
6. Antibodies to HIV and hepatitis C virus, the presence of the hepatitis B surface antigen, a positive syphilis test;
7. The presence of a sleep disorder (for example, night work, sleep disturbances, insomnia, recent return from another time zone, etc.);
8. Signs of alcohol or drug abuse; taking alcohol or drugs during 4 days before screening; smoking 3 months before screening;
9. History of allergies (including medicines and food products);
10. Blood donation / plasma, surgical intervention (in a hospital environment) during 12 weeks before screening;
11. Participation in other clinical trials or taking the study drug during 3 months before screening;
12. Acute infectious diseases less than 4 weeks before the start of the study;
13. Impossibility to understand or follow protocol instructions/

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events per treatment arm | Change from pre-dose to Day 28
  Adverse events have been classified according to CTCAE ver 4.03. Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version. For each preferred term, frequency counts and percentages will be calculated by cohort.The nature, severity, seriousness, and relationship to study medication will be summarized for all study subjects

SECONDARY OUTCOMES:
Pharmacokinetics of XC221GI by assessing AUC0-inf | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity
Pharmacokinetics of XC221A by assessing AUC0-inf | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity
Pharmacokinetics of XC221GI by assessing Cmax | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Maximum plasma concentration
Pharmacokinetics of XC221A by assessing Cmax | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Maximum plasma concentration
Pharmacokinetics of XC221GI by assessing AUC0-t | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of XC221A by assessing AUC0-t | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of XC221GI by assessing Tmax | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of XC221A by assessing Tmax | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of XC221GI by assessing T1/2 | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Terminal elimination half-life
Pharmacokinetics of XC221A by assessing T1/2 | Day 1 and 11 (Pre dose, 15 min, 30 min, 1,1.5, 2, 2.5, 3, 4, 5, 6, 8,12 and 16 h post dose), Day 2 and Day 12 (24 h ±10 min post dose), Day 3 and Day 13 (48 h ±10 min post dose), Day 4 and Day 14 (72 h ±10 min post dose), Day 7 to 10 (Pre dose)
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- SBEI HPE The First Moscow State Medical University n.a. Sechenov of Ministry of Health of Russian Federation, University Hospital #2, Department of Development of New Medicines, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No